CLINICAL TRIAL: NCT05399615
Title: Detection of Bacterial and Viral Pathogens Infection Among Hospitalized Patients Feasibility Study
Acronym: Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the company decision
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ID-PMC-2021
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-05

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospitalized Patients (Experimental): Patients hospitalized in internal ward at "Poriya" Medical Center
  Interventions: Diagnostic Test: VOX
- Controls (Experimental): Healthy volunteers
  Interventions: Diagnostic Test: VOX

INTERVENTIONS:
Diagnostic Test: VOX — Breath biopsy

SUMMARY:
Detection of bacterial and viral pathogens infection among hospitalized patients using breath analysis - feasibility study.

DETAILED DESCRIPTION:
A diagnostic prospective single-site study, with no anticipated risks or constraints.

Primary objective: To identify a set of breath Volatile Organic Compound biomarkers that enable the detection of pathogens infection and inflammatory response to pathogens infection among hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years at the time of consent
* Capable of understanding written and/or spoken language
* Able to provide informed consent
* Negative results for SARS-CoV-2
* Diagnosed with suspected respiratory infection

Exclusion Criteria:

* Under guardianship or deprived of liberty
* Pregnant or lactating woman
* Not able to breathe through mask for 8 minutes
* Intubated patients
* Patients in critical condition
* Diagnosed with hospital-acquired infection
* Medical history of malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Discovery of exhaled breath biomarkers | Through the study completion, up to 3 months.
  To evaluate the sensitivity, specificity, positive and negative predictive value of metabolomic biomarkers in exhaled breath samples as compared with pathogens biomarkers found in participants' blood and sputum samples.

SECONDARY OUTCOMES:
The association of exhaled biomarkers with inflammatory known biomarkers. | Through the study completion, up to 3 months.
  To measure the association between exhaled biomarkers and inflammatory known biomarkers that are found in participants' blood and sputum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Peretz, PhD, Principal Investigator — Poriya Medical Center
Locations (1):
- Poriya Medical Center, Poria – Neve Oved, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD